CLINICAL TRIAL: NCT05716542
Title: Prehabilitation to Revolutionize Oncology: Telehealth Exercise for Cognitive Triumphs (The PROTECT Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202302077
Record Dates: First submitted 2023-01-17; First posted 2023-02-08 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Cancer of the Breast
Keywords: prehabilitation; physical activity; cancer-related cognitive decline; telehealth; physical therapy; survivorship; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity Intervention (Experimental): * Participants will complete a primarily home-based PA intervention, with the goal of safely increasing their steps/day by incorporating moderate-to-vigorous physical activity (MVPA)
  * Participants will receive Fitbits with heart rate capabilities to support maintenance of the prescribed intensity during home exercise sessions and participants' self-monitoring of daily steps.
  * Participants will strategize aerobic MVPA behaviors with the intervention PT to identify preferable and enjoyable PA modalities (e.g., walking, cycling), while also identifying alternative options to allow for flexibility if life- or cancer-specific barriers arise
  * During the first Zoom coaching session, the intervention PT will train participants on using the Fitbit and completing home exercise logs. The PT will continue to meet with participants to support exercise maintenance, review home exercise sessions, strategize new exercises, and troubleshoot emerging chemotherapy-related health declines.
  Interventions: Other: Physical Activity Intervention
- Usual care, wait-list control condition (No Intervention): -Participants in the control group will proceed with their treatment regimen as prescribed by their oncologist(s). To prevent drop out and high attrition rates as well as promote healthy behavior, control group participants will receive a Fitbit at the initial set-up meeting to wear during chemotherapy, as well as an individualized home exercise program and up to two Zoom coaching sessions with a PT after chemotherapy completion.

INTERVENTIONS:
Other: Physical Activity Intervention — Fitbit wearable device, home exercise sessions, and telehealth appointments with physical therapist.
  Arms: Physical Activity Intervention

SUMMARY:
The investigators propose to deliver a pilot randomized controlled trial to 40 women newly diagnosed with breast cancer and scheduled to undergo chemotherapy. The current objectives are: 1) to evaluate the preliminary efficacy of the prehabilitation physical activity (PA) intervention delivered by a physical therapist and 2) assess the intervention's feasibility, acceptability, and appropriateness. The long-term goal is to scale this intervention for implementation into the standard of cancer care to prevent, mitigate, and treat cancer-related cognitive decline (CRCD).

ELIGIBILITY:
Eligibility Criteria:

* Diagnosis of breast cancer (stage I-III).
* Female.
* At least 18 years old.
* Scheduled to receive curative-intent chemotherapy.
* English speaking.
* Deemed fit to participate in a PA intervention by their oncologist.
* Not currently participating in another physical activity research study.
* Low active, defined by self-report as no more than 2 times per week of regular physical activity in the last six months
* Able to understand and willing to sign an IRB-approved written informed consent document.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Changes in self-reported cognition function as measured by FACT-Cog | Pre-chemotherapy and post-chemotherapy (estimated to be 12 weeks)
  The FACT-Cog examines a range of self-reported cognitive domains, including perceived cognitive impairment (PCI, range 0-71), perceived cognitive abilities (PCA, range 0-28), impact of cognitive impairment on quality of life (CogQOL, range 0-16), cognitive impairment perceived by others (CogOth, range 0-16), and a total cognitive functioning score (the sum of the other 4 subscales). Higher scores indicate fewer cognitive difficulties.
Feasibility of the intervention as measured by Feasibility of Intervention Measure (FIM) | After completion of intervention (estimated to be 12 weeks)
  The FIM measures the degree to which a participant feels an intervention is feasible to them. It ranges from 4-20, and higher scores indicate more feasibility. We will use a cutoff of 16 to indicate "feasible"

SECONDARY OUTCOMES:
Changes in objective measures of cognition function as measured by BrainBaseline Spatial Working Memory | Pre-chemotherapy and post-chemotherapy (estimated to be 12 weeks)
  BrainBaseline is a tool that delivers a battery of objective cognitive tests. The investigators will measure the participant's ability to hold information about an object's location in short term memory. Overall accuracy is the primary measure of performance. Accuracy ranges from 0-100%. Higher accuracy scores represent better accuracy.
Changes in objective measures of cognition function as measured by BrainBaseline N-back | Pre-chemotherapy and post-chemotherapy (estimated to be 12 weeks)
  BrainBaseline is a tool that delivers a battery of objective cognitive tests. The investigators will assess the participant's ability to retain sequentially presented information in short-term memory. Overall accuracy is considered the primary measure of performance.
  Accuracy ranges from 0-100%. Higher accuracy scores represent better accuracy.
Changes in objective measures of cognition function as measured by BrainBaseline Flanker | Pre-chemotherapy and post-chemotherapy (estimated to be 12 weeks)
  BrainBaseline is a tool that delivers a battery of objective cognitive tests. The investigators will assess the participant's ability to focus attention and block irrelevant information. Task performance is assessed by observing reaction time cost. Reaction time ranges from 0-5000 milliseconds. Higher reaction times represent slower reaction time.
Changes in objective measures of cognition function as measured by BrainBaseline Trails A&B | Pre-chemotherapy and post-chemotherapy (estimated to be 12 weeks)
  BrainBaseline is a tool that delivers a battery of objective cognitive tests. The investigators will assess the participant's ability to connect-the-dots, drawing a line between targets in a specified ascending order. Task performance is assessed by observing time to completion. A higher time to completion represents a slower ability to connect-the-dots.
Changes in objective measures of cognition function as measured by BrainBaseline Stroop | Pre-chemotherapy and post-chemotherapy (estimated to be 12 weeks)
  BrainBaseline is a tool that delivers a battery of objective cognitive tests. The investigators will measure the participant's ability to focus attention on a particular stimulus dimension while ignoring another. Task performance is assessed by observing the reaction time cost. Reaction time ranges from 0-5000 milliseconds. Higher reaction time scores represent slower reaction time.
Changes in objective measures of cognition function as measured by BrainBaseline Task switching | Pre-chemotherapy and post-chemotherapy (estimated to be 12 weeks)
  BrainBaseline is a tool that delivers a battery of objective cognitive tests. The investigators will measure the participant's ability to switch between two separate tasks. The primary outcome measure is switch cost. Reaction time ranges from 0-5000 milliseconds. Higher reaction time scores represent slower reaction time.
Changes in objective measures of cognition function as measured by BrainBaseline Digit Symbol Substitution | Pre-chemotherapy and post-chemotherapy (estimated to be 12 weeks)
  BrainBaseline is a tool that delivers a battery of objective cognitive tests. The investigators will measure the participant's ability to quickly and precisely shift attention from location to another, as well as measuring motor skill. The primary outcome measure is the number of correct substitutions made within the 90-second limit.
Acceptability of the intervention as measured by the Acceptability of Intervention Measure (AIM) | After completion of intervention (estimated to be 12 weeks)
  The AIM measures the degree to which a participant feels an intervention is acceptable to them. It ranges from 4-20, and higher scores indicate more acceptability. The investigators will use a cutoff of 16 to indicate "acceptable"
Appropriateness of the intervention as measured by the Intervention Appropriateness Measure (IAM) | After completion of intervention (estimated to be 12 weeks)
  The IAM measures the degree to which a participant feels an intervention is appropriate for them. It ranges from 4-20, and higher scores indicate more appropriateness. The investigators will use a cutoff of 16 to indicate "appropriate"
Adherence of the intervention as measured by percentage of home exercise sessions and PT telehealth appointments completed | After completion of intervention (estimated to be 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Peterson, M.D., MSCR, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu